CLINICAL TRIAL: NCT02713958
Title: The Efficacy of Telerehabilitation Program for Improvement of Upper Limb Function Among Adults Post Elbow Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Yafi Levanon PhD, Deputy of Occupational Therapy department, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-15-2296-RP-CTIL
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Elbow Fractures
Keywords: Telerehabilitation; Elbow fractures; Arthrolysis; MediTouch; Occupational Therapy; Active exercises
MeSH Terms: conditions — Elbow Fractures | interventions — Telerehabilitation; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tele rehabilitation (Experimental): Telerehabilitation:The subjects in the study group will receive two treatments in Telerehabilitation and one treatment in the clinic weekly . At home they will be asked practice daily active exercises with the Meditouch Ltd. system.
  Interventions: Other: Telerehabilitation
- rehabilitation (Active Comparator): Traditional Occupational Therapy:The subjects in this group will receive three treatments in the clinic every week. At home they will be asked to practice daily active exercises in the same level of difficulty and duration as the study group but without the Meditouch Ltd. system
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Telerehabilitation: Telerehabilitation treatment using a computerized system (MediTouch) for improving the elbow motion
  Arms: Tele rehabilitation
Other: Rehabilitation — Traditional Occupational Therapy treatment: Active exercises for elbow motion
  Arms: rehabilitation

SUMMARY:
This experimental research aims to examine the efficacy of Telerehabilitation treatment using a computerized system (MediTouch) in improving the upper limb function post elbow fractures. 24 participants aged 18-80 who are post surgery to fixate elbow fractures or arthrolysis of the elbow will be invited to participate in the study. The subjects will be matched into two groups according to age and fracture type to study and control groups. Both groups will be treated for a month in ambulatory clinic in the hospital and will do self-practice at home according to a intervention protocol. The subjects in the experimental group will receive two treatments in Telerehabilitation and one treatment in the clinic weekly, and the subjects in the control group will receive three treatments in the clinic every week. Activity daily living (ADL), Range of Motion, Hand strength disability and pain will be assessed before and after the intervention in order to asse the efficacy of the intervention.

DETAILED DESCRIPTION:
The elbow joint has an important role in the upper limb function. The rehabilitation process after injury is complex as a result of the common complications of the elbow after trauma, as stiffness, restriction in range of motion and occurrence of Heterotopic Ossification. According to the literature, early active mobilization reduces the incidence of these complications. Yet, current treatment protocols are based mainly on clinical experience and there is a lack in evidence-based trials regarding their efficiency. Recently, Occupational Therapists include Telerehabilitation in their treatments, using advanced technologies, which can be adapted to orthopedic injuries. The reported advantages of Telerehabilitation are the option to do self-practice without the need of arriving at a medical center and greater motivation to practice. This experimental research will examine the efficacy of Telerehabilitation treatment using a computerized system (MediTouch) in improving the upper limb function post elbow fractures.

This research will include 24 participants aged 18-80, from the hand surgery unit in Sheba medical center, who are post surgery to fixate elbow fractures or arthrolysis of the elbow, which is steady to mobilize. Patients diagnosed with rheumatology, neurological or orthopedic conditions and injuries in ligaments or nerves will be excluded. The subjects will be matched into two groups according to age and fracture type to study and control groups. Both groups will be treated for a month in ambulatory clinic in the hospital and will do self-practice at home. The subjects in the study group will receive two treatments in Telerehabilitation and one treatment in the clinic weekly, and the subjects in the control group will receive three treatments in the clinic every week. All subjects will be assessed before and after the intervention for hand function in everyday activities using The Jebsen-Taylor Hand Function Test, for disability and symptoms due to the injury using The Disabilities of the arm, shoulder and hand questionnaire, for pain and disability after injury in the elbow using The Patient-Rated Elbow Evaluation, for range of motion using Goniometer and for strength using Dynamometer. The Participants in the study group will also fill out questionnaires to evaluate level of satisfaction from the treatment and of the system usability. The hypotheses will be tested by the differences between groups in range of motion, function and satisfaction measures in order to assess the efficacy of the treatment in Telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Post surgery to fixate elbow fractures or arthrolysis of the elbow, which is steady to mobilize

Exclusion Criteria:

* Patients diagnosed with rheumatology, neurological or orthopedic conditions and injuries in ligaments or nerves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Range of motion | Change of range of motion in degrees from baseline up to 6 weeks

SECONDARY OUTCOMES:
The Disabilities of the arm, shoulder and hand questionnaire (Dash), | Change of Dash score from baseline up to 6 weeks
The Patient-Rated Elbow Evaluation (PREE) | Change of PREE score from baseline up to 6 weeks
Jebsen and Taylor functional test | Change of Jebsen score from baseline up to 6 weeks
Grip force | Change of grip force in kg from baseline up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ram Palti, Md, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No